CLINICAL TRIAL: NCT03898453
Title: EMDR Psychotherapy of Anxious-depressive Symptoms for Women That Present an Invasive Breast Cancer : a Randomised Controlled Trial
Brief Title: EMDR Psychotherapy for Anxious-depressive Symptoms in Breast Cancer Patient
Acronym: PSYCANCER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Régional Metz-Thionville (Other)
Collaborators: University of Lorraine (Other); Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2018-A01128-47
Record Dates: First submitted 2019-01-30; First posted 2019-04-02 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2022-09

CONDITIONS: Breast Cancer Female
Keywords: Breast Cancer; support psychotherapy; EMDR therapy; anxiety disorders
MeSH Terms: conditions — Breast Neoplasms; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Two groups assignment - One group will receive EMDR psychotherapy the other one support psychotherapy.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group EMDR psychotherapy (Experimental): Visit 0 : patient inclusion (questionnaires and interview) Visit 1 : anamnesis Visit 2 : patient stabilisation Visit 3 : EMDR psychotherapy care Visit 4 : EMDR psychotherapy care Visit 5 : EMDR psychotherapy care and questionnaires Visit 6 : EMDR psychotherapy care Visit 7 : EMDR psychotherapy care and questionnaires Follow-up 8 (three month after) : data recovery (questionnaires) Follow-up 9 (six month after) : data recovery (questionnaires)
  Interventions: Behavioral: EMDR psychotherapy
- Group Control : support psychotherapy (Other): Visit 0 : patient inclusion (questionnaires and interview) Visits 1-7: several methods could be used: psychoeducation about cancer and psychotherapy, positive interaction and activity schedule, emotional support , relaxation, prevention techniques… Questionnaires will be completed by patients at visit 5 and 7.
  Follow-up 8 (one month after) : data recovery (questionnaires) Follow-up 9 (six month after) : data recovery (questionnaires)
  Interventions: Behavioral: support psychotherapy

INTERVENTIONS:
Behavioral: EMDR psychotherapy — Visit 0 : patient inclusion (questionnaires and interview) Visit 1 : anamnesis Visit 2 : patient stabilisation Visit 3 : EMDR psychotherapy care Visit 4 : EMDR psychotherapy care Visit 5 : EMDR psychotherapy care and questionnaires Visit 6 : EMDR psychotherapy care Visit 7 : EMDR psychotherapy care and questionnaires Follow-up 8 (three month after) : data recovery (questionnaires) Follow-up 9 (six month after) : data recovery (questionnaires)
  Arms: Group EMDR psychotherapy
Behavioral: support psychotherapy — Visit 0 : patient inclusion (questionnaires and interview) Visits 1-7: several methods could be used: psychoeducation about cancer and psychotherapy, positive interaction and activity schedule, emotional support , relaxation, prevention techniques… Questionnaires will be completed by patients at visit 5 and 7.
  Follow-up 8 (one month after) : data recovery (questionnaires) Follow-up 9 (six month after) : data recovery (questionnaires)
  Arms: Group Control : support psychotherapy

SUMMARY:
The study will consist in an evaluation of the EMDR (Eye Movement Desensitization and Reprocessing) psychotherapy in the context on invasive primitive breast cancer. EMDR could then allow the affected patients to readjust their point of view on the pathology and thus promote more adapted behaviors or additional resources to cope with the disease. 190 Patients are going to be randomized in two groups : one group with EMDR psychotherapists and one group with support psychotherapists. Patients will receive 8 sessions. We expect that patient in EMDR psychotherapists group will have an higher decrease of anxiety score, depressive score (CES-D) and PTSD score, and a higher increase in quality of life.

DETAILED DESCRIPTION:
The study will consist in an evaluation of the EMDR psychotherapy in the context on invasive primitive breast cancer. EMDR could then allow the affected patients to readjust their point of view on the pathology and thus promote more adapted behaviors or additional resources to cope with the disease. 190 Patients are going to be randomized in two groups : one group with EMDR psychotherapists and one group with support psychotherapists. Patients will receive 8 sessions. We expect that patient in EMDR psychotherapists group will have an higher decrease of anxiety score, depressive score and PTSD score, and a higher increase in quality of life (QLQ)

ELIGIBILITY:
Inclusion Criteria:

* Being a 18 or more year old woman
* Having primary breast cancer or going to start treatment or having completed treatments for less than 6 months
* Presenting a state-anxiety level a score higher than 35.
* Being able to complete questionnaires.
* Having signed the consent letter
* Be affiliated to a social security system

Exclusion Criteria:

* Have contraindications for EMDR psychotherapy (neurological disorders, dissociative states, oculomotor problems)
* Have metastatic breast cancer
* physical multiple pathologies
* Have a psychiatric history (including anxio-depressive disorders). Background Assessment from M.I.N.I. (Sheehan et al., 1997)
* Present an addiction, an abuse of drugs or alcohol
* Person placed under the protection of justice, guardianship or trusteeship.
* Pregnant or lactating woman

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2019-03-11 (Actual); Primary Completion 2023-09-24 (Actual); Study Completion 2023-09-24 (Actual)

PRIMARY OUTCOMES:
State Anxiety | Month 9
  STAI-Y-A (State-Trait Anxiety Inventory) This questionnaire consists of a 20-items. The state version (STAI Y-A) indicate for 20 items and on 4-point Likert-Scale (not at all, somewhat, moderately so, and very much so) the extent to which they are currently experiencing each symptoms of anxiety. The total score ranges from 20 to 80. A higher total score indicate a higher level of anxiety.

SECONDARY OUTCOMES:
quality of life of cancer patients | Month 9
  EORTC QLQ-C30 Questionnaire The European Organization for research and Treatment of Cancer 30-item Quality of life (QoL) questionnaire is a well-validated health-related QoL instrument.
depression | Month 9
  CES-D (The Center for Epidemiologic Studies Depression) Questionnaire
posttraumatic symptoms | Month 9
  PTGI (The Posttraumatic Growth Inventory) Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Raffaele LONGO, Dr, Principal Investigator — CHR Metz-Thionville
Locations (1):
- CHR Metz-Thionville, Metz, France

IPD SHARING:
Plan to Share IPD: No